CLINICAL TRIAL: NCT04039191
Title: Short Messaging Service (SMS) Education for Post-operative Pain
Brief Title: SMS Education for Post-operative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Yufei Chen, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT2019-CHEN-SMS
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Opioid Use; Pain, Postoperative
Keywords: SMS; Education; Opioid Use; Pain; postoperative
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS survey (Placebo Comparator): Subject to receive SMS survey.
  Interventions: Behavioral: SMS survey
- SMS survey with education (Active Comparator): Subject to receive SMS survey with education.
  Interventions: Behavioral: SMS education

INTERVENTIONS:
Behavioral: SMS education — Patients will receive additional educational SMS messages post-operatively
  Arms: SMS survey with education
Behavioral: SMS survey — Patients will receive survey questions about post-operative pain and opioid use but no education
  Arms: SMS survey

SUMMARY:
The purpose the research is to assess whether or not postoperative education and awareness about pain and opioid use through SMS text messages will reduce overall opioid utilization after common outpatient surgeries.

DETAILED DESCRIPTION:
1.0 BACKGROUND, RATIONALE Since the turn of the century, opioid prescriptions and opioid-related overdose deaths in the United States has been on the rise, and is seen as the main cause of the consecutive decrease in life expectancy seen in 2015-2016. This epidemic has been declared a Public Health Emergency by the Department of Health and Human Services (HHS), with approximately 115 people dying daily from opioid-related drug overdoses nationwide. Over 40% of these overdoses are associated with prescription opioid abuse.

While non-medical opioid use is seen most commonly in those aged 15-24, accidental opioid overdose rates are highest in the those aged 45-54, an age group in which the medical use of opioids is most common. For many adults, their first medical exposure to opioids is following a surgical procedure. New persistent opioid use has been identified following both minor and major surgical procedures in 5.9% to 6.5% of patients, and was associated with behavioral and pain disorders rather than surgical pain itself. Furthermore, prolonged opioid use beyond 5 days, and even more so when the prescription exceeds 10 days, has been associated with an increased probability of continued long term opioid use.

Better pain management strategies and better research are key strategies the HHS have identified to combat the growing opioid epidemic. Current prescription patterns in the US are highly variable, although initiatives have been put into place to develop evidence based guidelines. Prescription opioid use has previously been linked to improved patient satisfaction with care, and in a study of primary care providers, those physicians who were incentivized by patient satisfaction scores reported an increased impact of these scores on their opioid prescribing practices. However, multiple studies have revealed no correlation between patient satisfaction scores and the amount of postoperative opioids prescribed.

A systematic review of studies describing opioid oversupply after surgery reported that 67-92% of patients reported unused opioids with few storing or disposing of excessive pills in an appropriate manner. Multiple studies have looked at interventions on the provider side, in order to minimize opioid prescriptions and thus minimize the availability of excess opioids that may facilitate opioid dependence and diversion into the community. While there has been an almost universal reduction in opioids prescribed, fewer studies have demonstrated a reduction in actual opioids taken by the patient.

Hill et al identified in 642 patients undergoing 5 common outpatient procedures a wide variation in the number of opioid pills prescribed and identified an ideal number of opioid pills per procedure that would adequate treat postoperative pain in the majority of patients, a number that was typically less than 50% of what was historically prescribed. The same group then presented their findings at their institution and recommended prescribers to encourage patients to use nonopioid analgesics. They found that following this education, there was a significant reduction in number of opioid pills prescribed across all procedures and also a decrease in the mean number of pills taken by patients following inguinal hernia and partial mastectomy with sentinel lymph node biopsy (SLNB) patients.

Howard et al reported a decrease in median amount of opioids prescribed for laparoscopic cholecystectomy from 250mg to 75mg following the development and education of physicians on evidence based prescribing guidelines. This was associated with no increase in the frequency of refill requests and a median postoperative opioid use reduction from 30mg to 20mg without a change in pain score. Similar results were seen in a group of oncology patients undergoing breast and melanoma procedures.

Several studies have also incorporated preoperative patient education about expected postoperative recovery and pain management strategies. However, most of these studies have been retrospectively performed in the context of quality improvement projects, with the comparison of preinterventional and postinterventional cohorts of patients.

Shindo et al in a retrospective cohort study of patients undergoing thyroid and parathyroid surgery reported a significant decrease in the amount of opioids prescribed following an intervention including preoperative patient counselling regarding pain management, the use of multimodality nonopioid pain management and the education of nurses and physicians. Prabhu et al took a shared decision-making approach to opioid prescribing utilizing a tablet computer based decision aid and found that patients who participated chose a 50% decreased in the number of opioids prescribed postoperatively.

Holman et al performed a retrospective cohort study on orthopedic trauma patients and found that patients who were instructed at the time of index procedure that they would receive prescription opioids for a maximum of 6 weeks were significantly more likely to have stopped using opioids by that time, although this effect was lost at 12 weeks.

Prospective studies evaluating the effects of these interventions have been fewer. Hartford et al developed a 4-pronged opioid intervention involving the implementation of patient education, healthcare provider education, intraoperative and postoperative multimodal analgesia with opioid reduction strategies in patients undergoing laparoscopic cholecystectomy or open hernia repair and evaluated their results prospectively. They found no difference in patient reported average postoperative pain scores but improvements in patient reported pain control. They also found a decrease in the number of opioids prescribed by the provider and ultimately filled by the patient.

Sugai et al randomized patients who underwent outpatient aesthetic surgery to preoperative education on how the body responds to pain and the side effects of opioids. Compared with patients who did not receive education in whom 100% filled their opioid prescription, they found that 90% of patients who received education declined a postoperative opioid prescription. Furthermore, patients in the control group had significantly greater postoperative average pain scores and a significantly longer duration of pain.

Alter et al performed a prospective randomized controlled trial of patients undergoing carpal tunnel release surgery and found that patients randomized to formal preoperative opioid counseling had reduced postoperative opioid consumption compared with patients without counselling (1.4 vs 4.2 opioid pills).

While preoperative patient education is undoubtedly useful, there is also an opportunity to monitor patients postoperatively and provide real-time feedback and reinforcement about pain management strategies and appropriate opioid use. The investigators have previously assessed real-time postoperative pain and opioid use in patients undergoing thyroid and parathyroid surgery utilizing a novel SMS survey (Chen et al, unpublished data). Overall response rate was >80% and the investigators were able to identify risk factors for patients who had prolonged opioid use, beyond what was expected after thyroid and parathyroid surgery. Although no intervention was performed in this study, it could potentially help identify patients in whom closer follow-up and earlier intervention might be beneficial.

The investigators theorize that real-time feedback and education about appropriate opioid use postoperatively may lead to a reduction in actual opioids consumed by the patient. The investigators propose a prospective randomized controlled trial to evaluate this in patients undergoing elective outpatient surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged ≥18 who are undergoing outpatient surgery (admission <23hrs) where opioids are typically prescribed

Exclusion Criteria:

* Non-English speaking patients.
* No access to cellphone.
* Admission beyond 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Number of opioid pills consumed | 10 days post-op
  Number of opioid pills consumed

SECONDARY OUTCOMES:
Post-operative pain scores | 10 days post-op
  Pain score will be utilizing a numeric pain rating scale (0-10) where 0 corresponds to no pain and 10 to worst pain.
  Total pain score will be reported as well as total scaled pain score which is total pain score divided by response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Yufei Chen, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States